CLINICAL TRIAL: NCT06224543
Title: Evaluate Artificial Intelligence (AI) Synthesized MR Images From Low Dose Gadobutrol CNS Images vs Standard Dose Gadobutrol CNS Images
Brief Title: MR Image Synthesis With Low Gadobutrol Dose and AI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Subtle Medical (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22403
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Enhancing Brain Lesions
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Intervention Model Description: Two interventional groups: Group A: 0.01 mmol/kg GV, Group B: 0.025 mmol/kg GV. Both groups also receive GV standard dose (0.1 mmol/kg) that serves as the clinical image set for the participant and as comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group A (10% dose GV) (Active Comparator): Each participant will receive a Standard dose gadobutrol (0.1 mmol/kg) in Period 1 and 10% dose gadobutrol (0.01 mmol/kg) in Period 2. During study Period 1, each participant will receive gadobutrol as a single intravenous (IV) administration at the standard dose for contrast-enhanced MRI followed by study Period 2 where a single IV low dose (10% dose) of gadobutrol will be administered. There will be a washout period of at least 72 hours but less than 15 days between the two periods. The individual study duration will therefore range from 4 to 15 days.
  Interventions: Device: SubtleGAD; Drug: Gadobutrol
- Group B (25% dose GV) (Active Comparator): Each participant will receive a Standard dose gadobutrol (0.1 mmol/kg) in Period 1 and Study Period 2: 25% dose gadobutrol (0.025 mmol/kg) in Period 2. During study Period 1, each participant will receive gadobutrol as a single intravenous (IV) administration at the standard dose for contrast-enhanced MRI followed by study Period 2 where a single IV low dose (25% dose) of gadobutrol will be administered. There will be a washout period of at least 72 hours but less than 15 days between the two periods. The individual study duration will therefore range from 4 to 15 days.
  Interventions: Device: SubtleGAD; Drug: Gadobutrol

INTERVENTIONS:
Device: SubtleGAD — SubtleGAD is an image processing software developed to enhance MR images acquired with low dose gadobutrol.
Drug: Gadobutrol — Gadavist is indicated for use with magnetic resonance imaging (MRI) in adult and pediatric patients including term neonates to detect and visualize areas with disrupted blood brain barrier and/or abnormal vascularity of the central nervous system.
  Other Names: Gadavist Injection

SUMMARY:
Study 22403 is a Phase 1 / Proof of Concept exploratory investigation to assess the non-inferiority of low dose gadobutrol and SubtleGAD™, a software medical device using an Artificial Intelligence (AI) deep learning-based method to enhance the contrast signal from images acquired with low dose administration of gadobutrol (GAD) contrast. The primary objective is to demonstrate noninferiority of synthesized Central Nervous System (CNS) magnetic resonance (MR) images for 1 or 2 different gadobutrol-enhanced low-dose groups (0.01mmol/kg, and0.025 mmol/kg) compared to gadobutrol-enhanced CNS MR images at a standard dose of 0.1 mmol/kg. This investigation is a prospective, randomized, open label, multi-center study with blinded reads in participants with known or highly suspected CNS pathology. There will be at least 60 participants enrolled (30 per study arm). SubtleGAD will be used as a post-processing tool, prior to blinded read assessment of MR images acquired in either arm of the study.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent at least 18 years of age and less than or equal to 89 years of age.
2. Have known or highly suspected brain lesions referred for contrast-enhanced MRI of the CNS.
3. Have an estimated glomerular filtration rate (eGFR) value ≥ 60 mL/min/1.73m^2.
4. Be fully informed about the study, including provisions of the Health Insurance Portability and Accountability Act (HIPAA) as applicable, and being capable and willing to consent to participate.

Exclusion Criteria:

1. Considered clinically unstable or has a concomitant/intercurrent condition that would not allow participation in the study.
2. Diagnoses of multiple sclerosis or other disease process that is expected to change its enhancement pattern in the time period of the follow-up.
3. Brain pathology or abnormalities that are not considered lesions.
4. Any contraindication for MRI procedure or gadobutrol administration.
5. Has severe cardiovascular disease.
6. Is expected or is scheduled to have a change in any treatment or procedure between the two study periods that may alter image comparability.
7. Is scheduled or is likely to require a biopsy or any interventional therapeutic procedure from the first study MRI up to 24 hours after the second study MRI.
8. Women currently lactating, pregnant, or planning on becoming pregnant during the study.
9. Women of childbearing potential with a positive urine pregnancy test within 24 hours before either gadobutrol administration.
10. Receipt of any gadolinium-based contrast agent <72 hours prior to the study MRIs.
11. Participants with acute kidney injury.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Compare enhancement of SubtleGAD in 10% dose and 25% dose gadobutrol MR images. | 4 to 15 days
  Compare enhancing lesions in gadobutrol-enhanced central nervous system (CNS) magnetic resonance imaging (MRI) low dose groups (0.01 mmol/kg, 0.025 mmol/kg), and standard dose (0.1 mmol/kg).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Central Illinois Radiological Associates; OSF St. Francis Hospital Peoria, Peoria, Illinois
  - UMass Chan Medical School, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Pennsylvania State University, State College, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No